CLINICAL TRIAL: NCT01561677
Title: Consequences of Obstructive Sleep Apnea Syndrome (OSAS) on the Outcome and the Survival After Ischemic Subtentorial Stroke. Impact of the Treatment With Continuous Positive Airway Pressure (CPAP)
Brief Title: Consequences of Obstructive Sleep Apnea Syndrome (OSAS) After Ischemic Subtentorial Stroke.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 8670
Record Dates: First submitted 2012-03-06; First posted 2012-03-23 (Estimated); Last update posted 2018-06-11 (Actual); Status verified 2018-06

CONDITIONS: Obstructive Sleep Apnea Syndrome; Brain Infarction
Keywords: obstructive sleep apnea; syndrome survival; ischemic stroke; continuous positive airway pressure; handicap
MeSH Terms: conditions — Sleep Apnea, Obstructive; Brain Infarction; Ischemic Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (5):
- apnea/hypopnea index (AHI<5 : no OSAS) (No Intervention)
- apnea/hypopnea index (5≥AHI<15 : mild OSAS) (No Intervention)
- apnea/hypopnea index (15≤AHI<30 :moderate OSAS) (No Intervention)
- apnea/hypopnea index ( AHI≥30 : severe OSAS treated). (Active Comparator): Treated with CPAP
  Interventions: Device: Continuous Positive Airway pressure-RESPIRONICS
- apnea/hypopnea index ( AHI≥30:severe OSAS untreated). (Sham Comparator): Treated with sham CPAP (placebo)
  Interventions: Device: Sham Continuous Positive Airway pressure-RESPIRONICS

INTERVENTIONS:
Device: Continuous Positive Airway pressure-RESPIRONICS — obstructive sleep apnea syndrome survival ischemic stroke continuous positive airway pressure handicap
  Arms: apnea/hypopnea index ( AHI≥30 : severe OSAS treated).
Device: Sham Continuous Positive Airway pressure-RESPIRONICS — inefficient Continuous Positivie Airway pressure
  Arms: apnea/hypopnea index ( AHI≥30:severe OSAS untreated).

SUMMARY:
Obstructive Sleep Apnea Syndrome (OSAS) is associated with stroke as a risk factor but little is known about the consequences of OSAS on the outcome and the survival after stroke. The aim of the investigators study is first to evaluate the outcome and the survival of patients with stroke depending of OSAS (presence and severity of OSAS) and second to compare the outcome and survival of patients with severe OSAS depending on the treatment of the syndrome with nocturnal continuous positive airway pressure. The investigators hypothesis is that OSAS is associated with worst survival and outcome and needs to be treated at the subacute phase of stroke.

DETAILED DESCRIPTION:
Objective : The aim of our study is to evaluate the consequences of obstructive sleep apnea syndrome on the functional outcome and the survival after an ischemic stroke and to measure the impact of the treatment with continuous positive airway pressure on the outcome of patients with severe obstructive sleep apnea syndrome.Patients and methods : We will prospectively explore by polysomnography, 300 consecutive patients hospitalized for an ischemic stroke in the stroke units of university hospitals at the sub acute phase after stroke (J15±4). 1) We will compare the functional outcome, the neurological impairment, the peripheral endothelial function, the continuous blood pressure measure on 24 hours recording, the quality of life and the survival at 3, 6 and 12 months in four groups of patients depending on their apnea/hypopnea index 2) In patients with severe obstructive sleep apnea syndrome, we will explore the impact on the functional outcome, the neurological impairment, and the survival at 3, 6 et 12 months of a treatment with continuous positive airway pressure (CPAP) randomly compared to a treatment with sham CPAP (non efficacious pressure) during 3 months. Conclusion : This study should allow us to evaluate the consequences of obstructive sleep apnea syndrome on the outcome and the survival after ischemic stroke and the impact and the tolerance of the treatment with continuous positive airway pressure in patients with severe obstructive sleep apnea syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Brain infarction confirmed by brain imaging

  * follow up possible
  * Severity at admission and at one week follow up:
* NIHSS ≥ 4 or- isolated aphasia (item 9 ofNIHSS ≥ 1) or
* negligence (item 11 du NIHSS ≥ 2) or
* distal motor deficit (score ≥ 1)

  * Health insurance affiliation
  * Inform and free consent agreement

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2011-09 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
functional independence scale | 3 months
  The variation of the functional independence scale is evaluated by the Barthel Index at three months after stroke in four groups of patients depending on their apnea/hypopnea.In the patients group severe OSAS treated with CPAP from day 15 after stroke compared to patients with severe OSAS treated with sham CPAPThe neurological dependency will be evaluated by the Barthel Index .This scale measures the consequences of the motor and cognitive disorders on the daily living with 10 items.

SECONDARY OUTCOMES:
neurological impairment | 3 months
  The variation of the neurological impairment (NIHSS score) at three months after stroke:
  * in four groups of patients depending on their apnea/hypopnea index
  * In the patients group with severe OSAS treated with CPAP from day 15 after stroke vs patients with severe OSAS treated with sham CPAP
the handicap | 3 months
  the handicap (via the Rankin score ), at three months after stroke:
  in four groups of patients depending on their apnea/hypopnea index In the patients group with severe OSAS treated with CPAP from day 15 after stroke vs patients with severe OSAS treated with sham CPAP
blood pressure | 3 months
  The continuous measure of blood pressure over 24 hours at three months after stroke:
  in four groups of patients depending on their apnea/hypopnea index In the patients group with severe OSAS treated with CPAP from day 15 after stroke vs patients with severe OSAS treated with sham CPAP
the quality of life | 3 months
  the quality of life (SF-36) at three months after stroke:
  in four groups of patients depending on their apnea/hypopnea index In the patients group with severe OSAS treated with CPAP from day 15 after stroke vs patients with severe OSAS treated with sham CPAP
the survival | 3 months
  the survival at three months after stroke:
  in four groups of patients depending on their apnea/hypopnea index In the patients group with severe OSAS treated with CPAP from day 15 after stroke vs patients with severe OSAS treated with sham CPAP

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Montpellier, Montpellier, France

REFERENCES:
- [Derived] Denis C, Jaussent I, Guiraud L, Mestejanot C, Arquizan C, Mourand I, Chenini S, Abril B, Wacongne A, Tamisier R, Baillieul S, Pepin JL, Barateau L, Dauvilliers Y. Functional recovery after ischemic stroke: Impact of different sleep health parameters. J Sleep Res. 2024 Feb;33(1):e13964. doi: 10.1111/jsr.13964. Epub 2023 Jun 20. PMID 37338010